Official Study Title: Investigation of the Effect of Elastic Lower Extremity Orthosis on Gait and Balance Parameters in Children With Spastic Cerebral Palsy: A Randomized Controlled Trial

ClinicalTrials.gov Identifier: NCT07122362

**Document Date:** April 19, 2025

## **Statistical Analysis Plan (SAP)**

Analyses will be performed using IBM SPSS Statistics 26.0

Normality assessment: histograms, probability plots, Shapiro–Wilk test, skewness/kurtosis, coefficient of variation

Descriptive statistics: nominal/ordinal  $\rightarrow$  frequencies and percentages, numerical  $\rightarrow$  median  $\pm$  percentiles or mean  $\pm$  SD

Categorical variables: Chi-square (Pearson or Fisher)

Within-group comparisons (pre/post): Paired t-test / Wilcoxon

Between-group comparisons: Student t-test / Mann-Whitney U

Significance level: p < 0.05